CLINICAL TRIAL: NCT02430116
Title: Mitochondrial Apoptotic Pathway Induced by Myocardial Ischemia-Reperfusion Injury in Human
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: WANG Yan-bin (Other)
Responsible Party: Sponsor-Investigator, WANG Yan-bin, Clinical Professor, Shenzhen Sun Yat-sen Cardiovascular Hospital
Organization: Shenzhen Sun Yat-sen Cardiovascular Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: wangyanbin123
Record Dates: First submitted 2015-04-20; First posted 2015-04-30 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Ischemia-reperfusion(I/R); Cardiopulmonarybypass; the Mitochondrial Pathway; Ischemic Postconditioning
MeSH Terms: interventions — Ischemic Postconditioning

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- negative control group (No Intervention): The myocardial tissues of the right atrial appendage were obtained at 3 min before CPB was established in the NEG group.
- I/R group (Active Comparator): The myocardial tissues of the right atrial appendage were obtained at 45 min after opening the aorta in the I/R group.
  Interventions: Procedure: Ischemic postconditioning
- I-postC group (Experimental): The procedure involved 5 min before opening the ascending aorta, aortic unclamping for 30 s, and cross-clamping for 30 s for three cycles, after which the ascending aorta was completely opened.
  Interventions: Procedure: Ischemic postconditioning

INTERVENTIONS:
Procedure: Ischemic postconditioning — In the Treat group, the procedure involved 5 min before opening the ascending aorta, aortic unclamping for 30 s, and cross-clamping for 30 s for three cycles, after which the ascending aorta was completely opened.
  Other Names: The intervention is neither a drug nor a device. It is a procedure.
  Arms: I-postC group; I/R group

SUMMARY:
Background: The cardiomyocytes apoptosis induced by ischemia-reperfusion(I/R) is one of the most important factors in the myocardial I/R injury(MIRI) undergoing cardiac valve replacement with cardiopulmonary bypass(CVRCPB),and Ischemic postconditioning (I-postC) can inhibit apoptosis of myocardial cells. Consequently, this study investigated the key genes and apoptosis signaling pathways of myocardium in patients undergoing CVRCPB.

Methods: A total of 36 New York Heart Association class II or III patients with rheumatic heart disease (RHD) of both sexes, aged 21-59 years, who were scheduled for first cardiac valve replacement with CPB in the investigators' hospital from February 2014 to May 2015, were randomly divided into the following three groups (n=12 each): negative control group (NEG group); I/R group (POS group); and I-postC group (Treat group). In the Treat group, the procedure involved 5 min before opening the ascending aorta, aortic unclamping for 30 s, and cross-clamping for 30 s for three cycles, after which the ascending aorta was completely opened. The NEG and Treat groups were not treated. Thirty-six patients were assessed for arrhythmia and recovery of myocardial contractile function after reperfusion by electrocardiograms and degree of dependence on vasoactive drugs. The myocardial tissues of the right atrial appendage were obtained at 3 min before CPB was established in the NEG group, and at 45 min after opening the aorta in the POS and Treat groups. In all three groups, the myocardial tissues of the right atrial appendage were obtained and preserved at -80°C for further experiments. The right atrial appendage of three patients randomly selected in each group was fixed with RNA later (Qiagen, Hilden, Germany) in a centrifuge tube overnight at 4°C, and then preserved at -20°C for RNA extraction. Human 12×135K Gene Array profiling of mRNA expressions was undertaken in human cardiac muscle cells. Differentially expressed mRNAs verified by quantitative real-time RT-PCR were subjected to pathway analysis. The mRNA expressions of AIF, APAF1, CYCS, Bax, caspase-3, caspase-9, caspase-6, caspase-7, BCL2, BAG1, and PI3K were assessed by real-time RT-PCR and western blot analysis. The levels of myocardial apoptosis induced by I/R were investigated by TUNEL assays. The changes in MIRI induced by myocardial apoptosis were investigated by pathologic examination of the myocardium.

ELIGIBILITY:
Inclusion Criteria:

* New York Heart Association class II or III
* aged 21-59 years
* scheduled for first cardiac valve replacement with CPB

Exclusion Criteria:

* The patient with a history of heart operation or diabetes,
* with a history of liver and/or kidney dysfunction,
* with a history of coronary heart disease and the left ventricular ejection fraction(LVEF)<0.4, receiving drugs with pretreatment effectssuchas hormones, ATP-sensitive potassium (KATP) channel openers，insulin，et al. within preoperative one week,

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
recovery of myocardial contractile function after reperfusion | 1 day
degree of dependence on vasoactive drugs | 1 day
number of participants with postoperative arrhythmia | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen SUN Yat-Sen Cardiovascular hospital, Shenzhen, China